CLINICAL TRIAL: NCT02961114
Title: Use of Autologous Adipose-Derived Stem/Stromal Cells In Symptomatic Benign Prostate Hypertrophy
Brief Title: Use of Autologous Adipose-Derived Stem/Stromal Cells (AD-cSVF) in Symptomatic Benign Prostate Hypertrophy
Acronym: SVF-BPN
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID restrictions prevent patient enrollment or treatment. Clinical Trial facility is being closed due to viral limitations and loss of staff to perform
Sponsor: Robert W. Alexander, MD, FICS (Industry)
Collaborators: Terry, Glenn C., M.D. (Individual)
Responsible Party: Sponsor-Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Science, Healeon Medical Inc
Organization: Healeon Medical Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGV GARM 4
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: BPH; Nocturia; BPH With Urinary Obstruction; Prostatism; Prostate Inflammation
Keywords: Prostatitis, Chronic; Nocturia; BPH With Urinary Obstruction
MeSH Terms: conditions — Nocturia; Prostatism; Prostatitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Microcannula Harvest Adipose (Experimental): Acquisition of AD-tSVF via closed syringe microcannula harvest from subdermal fat deposits
  Interventions: Procedure: Microcannula Harvest Adipose
- Centricyte 1000 (Experimental): Autologous AD-tSVF via enzymatic isolation/concentration via Centricyte 1000 closed system to create AD-cSVF
  Interventions: Device: Centricyte 1000
- IV Sterile Normal Saline (Experimental): Re-suspension of AD-cSVF pellet in Normal Saline for deployment via IV
  Interventions: Biological: IV Sterile Normal Saline

INTERVENTIONS:
Procedure: Microcannula Harvest Adipose — Use of closed syringe microcannula harvest of autologous AD-tSVF from subdermal adipose deposits to create a AD-cSVF
  Arms: Microcannula Harvest Adipose
Device: Centricyte 1000 — Use of Centricyte 1000 closed system digestion, incubation/agitation, and centrifugation to acquire a concentrated pellet of AD-cSVF
  Arms: Centricyte 1000
Biological: IV Sterile Normal Saline — Sterile Normal Saline deployment of AD-cSVF in suspension of 500cc in IV pathway
  Arms: IV Sterile Normal Saline

SUMMARY:
Benign prostate hypertrophy (BPH) and inflammation are common non-cancerous enlargement of the prostate, which result in urinary interference and incomplete drainage of the bladder. Compression of the urethra is common cause of such resistance of full draining, and may over time result in progressive hypertrophy, instability, urgency, nocturia and weakness of the bladder musculature.

Prostatic growth frequently begins in the 30s, and it is estimated that 50% of all males have benign enlargement leading to 75% by age 80. BPH and low grade inflammation is one of the ten most prominent and costly disorders in males over 50.

Urinary tract symptoms are divided into issues of storage, voiding, and post-void symptoms can be associated with bladder outlet obstruction (BOO).

This study utilizes isolation of adipose-derived stem/stromal cellular stromal vascular fraction (AD-cSVF) deployed as an IV suspension in sterile Normal Saline (500cc). Due to the anti-inflammatory and immunomodulatory effects common to AD-cSVF are tested in relief of the inflammatory elements and the concurrent hypertrophy in BPH. Early pilot use has suggested a positive effect on these issues, and have relieved much of the incomplete voiding, pain, nocturia, delay in starting/stopping urination, and increased urgency and frequency.

Lipoharvesting of Adipose-Derived tissue stromal vascular fraction (AD-tSVF) is now a common closed access to subdermal adipose stromal/stem cell population consisting of both stem and stromal cells, each of which are felt to contribute a wide variety of effects and potentials. Closed, sterile isolation of the AD-cSVF is possible with advent of closed systems to enzymatically release these cells from the actual matrix (scaffolding) within the adipose tissue complex (ATC). This group of largely un-designated cell population is isolated and concentrated via a standard gradient layer separation by centrifugation. This cellular isolate is then suspended in an IV of 500 cc Normal Saline and reintroduced to the patient.

This study is examining the clinical safety and efficacy of this approach, as well as tracking the duration of effects and establish a therapeutic interval.

DETAILED DESCRIPTION:
Benign prostate hypertrophy (BPH) and inflammation are common non-cancerous enlargement of the prostate, which result in urinary interference and incomplete drainage of the bladder. Compression of the urethra is common cause of such resistance of full draining, and may over time result in progressive hypertrophy, instability, urgency, nocturia and weakness of the bladder musculature.

Prostatic growth frequently begins in the 30s, and it is estimated that 50% of all males have benign enlargement leading to 75% by age 80. BPH and low grade inflammation is one of the ten most prominent and costly disorders in males over 50. BPH is often a progressive disease and may lead to increased urinary stasis and increased risk of urinary tract infections.

Urinary tract symptoms are divided into issues of storage, voiding, and post-void symptoms can be associated with bladder outlet obstruction (BOO). Storage symptoms include need to urinate frequently, waking at night to urinate (nocturia), and incontinence (involuntary). Voiding issues include urinary hesitancy, intermittency (start/stopping flow), leaking after voiding and may include some pain (dysuria) associated with urination. Post-voiding symptoms include abdominal pain, feeling of full bladder, acute urinary retention and frequency, dysuria, hesitancy, etc.

Causation may be associated with age related changes in androgens (such as testosterone and others), but do not seem to be the direct cause of the enlargement.

Androgens promote prostate cell proliferation, but relatively low levels of testosterone are often found in patients with BPH.

Treatment often has been aimed at lifestyle change (exercise, decrease nighttime fluid intake, moderating alcohol and caffeine, decrease certain anticholinergic medications. Use of medication have some advantages, including alpha blocker and 5 alpha-reductase inhibitors, and some broad spectrum antibiotics (like Ciprofloxacin) seem to help many of those with increasing symptoms. Self catheterization and surgery are occasionally needed for patient comfort and reduction of symptomatology.

Alternative remedies include herbal remedies (saw palmetto) and anecdotal effects in patients receiving parenteral stem/stromal cell therapies for other clinical issues. Initially commented that the patient reported improvement of symptoms, have led to this study to determine if any long-interval therapy may be as effective as surgery or catheterization.

This study utilizes isolation of adipose-derived stem/stromal cellular stromal vascular fraction (AD-cSVF) deployed as an IV suspension in sterile Normal Saline (500cc). Due to the anti-inflammatory and immunomodulatory effects common to AD-cSVF are tested in relief of the inflammatory elements and the concurrent hypertrophy in BPH. Early pilot use has suggested a positive effect on these issues, and have relieved much of the incomplete voiding, pain, nocturia, delay in starting/stopping urination, and increased urgency and frequency.

Lipoharvesting of Adipose-Derived tissue stromal vascular fraction (AD-tSVF) is now a common closed access to subdermal adipose stromal/stem cell population consisting of both stem and stromal cells, each of which are felt to contribute a wide variety of effects and potentials. Closed, sterile isolation of the AD-cSVF is possible with advent of closed systems to enzymatically release these cells from the actual matrix (scaffolding) within the adipose tissue complex (ATC). This group of largely un-designated cell population is isolated and concentrated via a standard gradient layer separation by centrifugation. This cellular isolate is then suspended in an IV of 500 cc Normal Saline and reintroduced to the patient.

This study is examining the clinical safety and efficacy of this approach, as well as tracking the duration of effects and establish a therapeutic interval.

ELIGIBILITY:
Inclusion Criteria:

* Documented history BPH for at least 1 year
* AUA SI greater than or equal to score of 15
* Qmax < 15 ml/sec
* Severe nocturia
* Prostate Specific Antigen (PSA) > 4 ng/mL with documentation of non-malignancy

Exclusion Criteria:

* History of illness or conditions that may interfere with study or endanger subject
* Use of prescription medication that may interfere with study or endanger subject within 30 days
* History of surgical procedures for BPH or documented prostate cancer
* Post-void residual urine volumes of > 350 cc
* PSA > 10 ng/mL
* Prostate cancer not ruled out by biopsy if PSA is consistently higher than 4 ng/mL

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | Outcome measured at 1 month
  Report of minor and severe adverse effects caused by the procedures
Clinical Symptom Changes | Baseline, 1 Month, 6 Months, 1 years
  Assessment of change from baseline (0) of frequency, urgency, pain, voiding time, and flow rate during voiding

SECONDARY OUTCOMES:
Pain on Voiding | Baseline, 6 month, 1 year
  Visual Analog Pain Scale (VAS) designated as levels pain 1-10
Change of BPH Symptom Score | Baseline, 6 month, 12 month
  BPH Symptom Score change from baseline use American Urological Association Symptom Score Index change from baseline using Amercian Urological Association Symptom Score Index (AUA SI)
Change in BPH Symptom Score | Baseline, 6 month, 1 year
  Change from Baseline of Measured International Prostate Symptom Score (I-PPS)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Global Alliance for Regenerative Medicine-USA, Stevensville, Montana
  - Regenevita LLC, Stevensville, Montana

IPD SHARING:
Plan to Share IPD: Yes
Annual Data Update to All Collaborators

REFERENCES:
- [Background] Chang RT, Kirby R, Challacombe BJ. Is there a link between BPH and prostate cancer? Practitioner. 2012 Apr;256(1750):13-6, 2. PMID 22792684
- [Background] Guess HA, Arrighi HM, Metter EJ, Fozard JL. Cumulative prevalence of prostatism matches the autopsy prevalence of benign prostatic hyperplasia. Prostate. 1990;17(3):241-6. doi: 10.1002/pros.2990170308. PMID 1700403
- [Background] Fenter TC, Naslund MJ, Shah MB, Eaddy MT, Black L. The cost of treating the 10 most prevalent diseases in men 50 years of age or older. Am J Manag Care. 2006 Mar;12(4 Suppl):S90-8. PMID 16551207
- [Background] White JM JR, O'Brien DP III. Incontinence and Stream Abnormalities. In: Walker HK, Hall WD, Hurst JW, editors. Clinical Methods: The History, Physical, and Laboratory Examinations. 3rd edition. Boston: Butterworths; 1990. Chapter 185. Available from http://www.ncbi.nlm.nih.gov/books/NBK295/ PMID 21250138
- [Background] Sarma AV, Wei JT. Clinical practice. Benign prostatic hyperplasia and lower urinary tract symptoms. N Engl J Med. 2012 Jul 19;367(3):248-57. doi: 10.1056/NEJMcp1106637. No abstract available. PMID 22808960
- [Background] Bartsch G, Rittmaster RS, Klocker H. Dihydrotestosterone and the concept of 5alpha-reductase inhibition in human benign prostatic hyperplasia. World J Urol. 2002 Apr;19(6):413-25. doi: 10.1007/s00345-002-0248-5. PMID 12022710
- [Background] Lagiou P, Mantzoros CS, Tzonou A, Signorello LB, Lipworth L, Trichopoulos D. Serum steroids in relation to benign prostatic hyperplasia. Oncology. 1997 Nov-Dec;54(6):497-501. doi: 10.1159/000227609. PMID 9394847
- [Background] Roberts RO, Jacobson DJ, Rhodes T, Klee GG, Leiber MM, Jacobsen SJ. Serum sex hormones and measures of benign prostatic hyperplasia. Prostate. 2004 Oct 1;61(2):124-31. doi: 10.1002/pros.20080. PMID 15305335
- [Background] Ho CK, Nanda J, Chapman KE, Habib FK. Oestrogen and benign prostatic hyperplasia: effects on stromal cell proliferation and local formation from androgen. J Endocrinol. 2008 Jun;197(3):483-91. doi: 10.1677/JOE-07-0470. PMID 18492814
- [Background] Niu YJ, Ma TX, Zhang J, Xu Y, Han RF, Sun G. Androgen and prostatic stroma. Asian J Androl. 2003 Mar;5(1):19-26. PMID 12646998
- [Background] Chyou PH, Nomura AM, Stemmermann GN, Hankin JH. A prospective study of alcohol, diet, and other lifestyle factors in relation to obstructive uropathy. Prostate. 1993;22(3):253-64. doi: 10.1002/pros.2990220308. PMID 7683816
- [Background] Wasserman NF. Benign prostatic hyperplasia: a review and ultrasound classification. Radiol Clin North Am. 2006 Sep;44(5):689-710, viii. doi: 10.1016/j.rcl.2006.07.005. PMID 17030221
- [Background] Parsons JK. Benign Prostatic Hyperplasia and Male Lower Urinary Tract Symptoms: Epidemiology and Risk Factors. Curr Bladder Dysfunct Rep. 2010 Dec;5(4):212-218. doi: 10.1007/s11884-010-0067-2. Epub 2010 Sep 7. PMID 21475707
- [Background] Silva J, Silva CM, Cruz F. Current medical treatment of lower urinary tract symptoms/BPH: do we have a standard? Curr Opin Urol. 2014 Jan;24(1):21-8. doi: 10.1097/MOU.0000000000000007. PMID 24231531
- [Background] Roehrborn CG, Boyle P, Nickel JC, Hoefner K, Andriole G; ARIA3001 ARIA3002 and ARIA3003 Study Investigators. Efficacy and safety of a dual inhibitor of 5-alpha-reductase types 1 and 2 (dutasteride) in men with benign prostatic hyperplasia. Urology. 2002 Sep;60(3):434-41. doi: 10.1016/s0090-4295(02)01905-2. PMID 12350480
- [Background] Roehrborn CG, Bruskewitz R, Nickel JC, McConnell JD, Saltzman B, Gittelman MC, Malek GH, Gottesman JE, Suryawanshi S, Drisko J, Meehan A, Waldstreicher J; Proscar Long-Term Efficacy and Safety Study Group. Sustained decrease in incidence of acute urinary retention and surgery with finasteride for 6 years in men with benign prostatic hyperplasia. J Urol. 2004 Mar;171(3):1194-8. doi: 10.1097/01.ju.0000112918.74410.94. PMID 14767299
- [Background] Greco KA, McVary KT. The role of combination medical therapy in benign prostatic hyperplasia. Int J Impot Res. 2008 Dec;20 Suppl 3:S33-43. doi: 10.1038/ijir.2008.51. PMID 19002123
- [Background] Prieto J, Murphy CL, Moore KN, Fader M. Intermittent catheterisation for long-term bladder management. Cochrane Database Syst Rev. 2014 Sep 10;(9):CD006008. doi: 10.1002/14651858.CD006008.pub3. PMID 25208303
- [Background] Bent S, Kane C, Shinohara K, Neuhaus J, Hudes ES, Goldberg H, Avins AL. Saw palmetto for benign prostatic hyperplasia. N Engl J Med. 2006 Feb 9;354(6):557-66. doi: 10.1056/NEJMoa053085. PMID 16467543
- [Background] Ma CH, Lin WL, Lui SL, Cai XY, Wong VT, Ziea E, Zhang ZJ. Efficacy and safety of Chinese herbal medicine for benign prostatic hyperplasia: systematic review of randomized controlled trials. Asian J Androl. 2013 Jul;15(4):471-82. doi: 10.1038/aja.2012.173. Epub 2013 Jun 3. PMID 23728585